CLINICAL TRIAL: NCT04315857
Title: Pilot Study on Glycemic Variations in Diabetic Patients Treated With Chemotherapy: Benefit of Continuous Interstitial Glucose Measurement
Brief Title: Study on Glycemic Variations in Diabetic Patients Treated With Chemotherapy: Benefit of Continuous Interstitial Glucose Measurement
Acronym: ONCODIAB
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: PETIT 2019
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Diabetes; Chemotherapy; Interstitial Glycemia; Freestyle
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diabetics: diabetics receiving chemotherapy for cancer
  Interventions: Other: interstitial glycaemia

INTERVENTIONS:
Other: interstitial glycaemia — Continuous measurement of interstitial blood glucose during the first 15 days of the first two chemotherapy courses.

SUMMARY:
Over the last years, there has been a progressive increase in the prevalence of diabetes. Approximately 3.3 million French adults and approximately 425 million adults worldwide have been diagnosed with diabetes. Because of the associated high morbiditiy and mortality, this chronic disease is at the heart of public health discussions, and technologies to improve its management are constantly progressing.

One notable innovation is the Freestyle Free blood glucose meter, which enables the continuous measurement of interstitial blood glucose levels. This type of device has enabled diabetic patients to refine their blood glucose monitoring and improve the balance of their diabetes, while reducing the associated constraints.

To date, the Freestyle Libre meter is only available in patients treated with insulin pumps or multi-injections (at least 3 insulin injections per day) due to the risk of significant blood glucose variations. However, one can imagine other situations where the Freestyle Libre could be of interest to detect significant glycemic imbalances, such as in diabetic patients with cancer treated with chemotherapy.

To our knowledge, no study has been conducted on the relationship between chemotherapy and glycemic balance.

A few studies have looked at the balance of diabetes and chemotherapy in combination with corticosteroid therapy, but the analyses were based on fasting blood glucose levels, or some capillary blood glucose levels, or glycated hemoglobin - which can be deficient due to toxic treatments at the bone marrow level with variations in erythropoiesis. Hypoglycemia facilitated by anorexia (related to cancer and chemotherapy) or hyperglycemia facilitated by hyperglycemic drugs can be severe for patients with high care utilization and associated significant cost.

However, other studies have looked at the consequences of unbalanced diabetes in the context of cancer treated with chemotherapy. The results showed that hyperglycemia could lead to an increased risk of toxicity and side effects of chemotherapy. In addition, the choice of chemotherapy type or dosage may be different from a non-diabetic patient, which may result in a reduced remission and/or cure rate.

These results are then in contradiction with common practice, as the presence of cancer often leads doctors to be less rigorous in controlling blood sugar levels.

As the prevalence of diabetes in patients newly diagnosed with cancer is quite high (between 8 and 18% depending on the study) and because it is likely to continue to increase with the increasing prevalence of diabetes, particularly type 2 diabetes, closer monitoring of blood glucose levels in diabetic patients appears to be essential in the overall management of the patient.

In our study, we therefore focused on the continuous interstitial glycemia of diabetic patients entering the Ambulatory Medical Unit of Cancerology to start chemotherapy related to their cancer, be it hematological, digestive, cutaneous or gynecological.

ELIGIBILITY:
Inclusion Criteria:

* Person who has provided oral consent
* Diabetic cancer patient starting chemotherapy for the first time or after a period of remission of at least 6 months.

Exclusion Criteria:

* Person not affiliated to French National Health Insurance
* Person subject to legal protection (guardianship, trusteeship)
* Person subject to partial justice safeguard measure
* Pregnant, parturient or breastfeeding woman
* Adult unable to provide consent
* Minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patients starting chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Time spent with an interstitial blood glucose level below 0.70 g/l and above 2.5 g/l | Through study completion, an average of 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Legris P, Bouillet B, Paris J, Pistre P, Devaux M, Bost S, Simoneau I, Manfredi S, Drouillard A, Bastie JN, Chaix M, Massoud P, Rouland A, Aho S, Boulin M, Petit JM. Glycemic control in people with diabetes treated with cancer chemotherapy: contribution of continuous glucose monitoring. Acta Diabetol. 2023 Apr;60(4):545-552. doi: 10.1007/s00592-023-02032-z. Epub 2023 Jan 13. PMID 36637528